CLINICAL TRIAL: NCT03861598
Title: A Feasibility Study: Evaluating Carvedilol With Chemotherapy in Second Line Glioblastoma Multiforme and Response of Peripheral Glioma Circulating Tumor Cells
Brief Title: Carvedilol With Chemotherapy in Second Line Glioblastoma and Response of Circulating Tumor Cells
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Due to Covid
Sponsor: West Virginia University (Other)
Collaborators: West Virginia Clinical and Translational Science Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WVU010318
Record Dates: First submitted 2019-02-11; First posted 2019-03-04 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Glioblastoma Multiforme; Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort 1 (Experimental): Carvedilol orally with standard chemotherapy starting at 6.25 mg and increasing to 12.5 mg if tolerated after 1-2 weeks for a total of 4 cycles of treatment.
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — Carvedilol orally starting at 6.25 mg and increasing to 12.5 mg if tolerated after 1-2 weeks for a total of 4 cycles of treatment.
  Other Names: Coreg; Coreg CR

SUMMARY:
Subjects will receive standard chemotherapy and Tumor Treated Fields (TTFields) and will also receive Carvedilol for 4 cycles of treatment. Carvedilol will start at 6.25 mg orally twice a day and be increased to 12.5 mg orally twice daily after 1 to 2 weeks if tolerated. Peripheral glioma circulating tumor cells (CTC) and brain MRI with and without contrast will be obtained at baseline, 2 cycles, and 4 cycles to determine the efficacy and direction of change of the CTC using a new assay tool. Preliminary assessment of the tolerability of Carvedilol with standard chemotherapy will also be evaluated.

DETAILED DESCRIPTION:
This will be a feasibility study to assess the use of a new PCR assay with response to standard chemotherapy treatment in the second line setting in glioblastoma multiforme (GBM). The change in direction with the combination of carvedilol with standard of chemotherapy based upon brain MRI results will be assessed and associating that with also the change in the quantity of tumor cells with a new invented assay device. Six subjects will be enrolled in the study who have recurrent GBM and will be receiving second line treatment.

The subjects will receive standard therapy per the discretion of the treating oncologist. Carvedilol will start at 6.25 mg orally twice daily for 1-2 weeks to confirm tolerance. The subjects will then receive carvedilol at 12.5 mg orally twice daily as the maximum dose and take it continuously for 4 cycles of therapy. At the completion of 4 cycles, patients will stop taking carvedilol. If the patients were on previous anti-hypertensive medications, they will be instructed to restart those medications if stopped on this trial for carvedilol.

Peripheral blood samples will be collected at baseline before initiation of treatment, on first day of every cycle for four cycles and after the last cycle is completed to obtain peripheral glioma circulating tumor levels. Subjects will be re-evaluated for response every 2 cycles of therapy with brain MRI with and without contrast.

ELIGIBILITY:
Inclusion Criteria:

* Grade IV Glioblastoma, receiving chemotherapy with or without TTfields.
* Progressive or recurrent disease requiring second line treatment
* evidence of progression of disease by brain MRI and are planned to receive chemotherapy

Exclusion Criteria:

* Current use of another beta blocker that cannot be switched to carvedilol at the onset of the trial.
* Systolic blood pressure <90 mmHg and/or heart rate <60 bpm without hypertensive medications
* Allergy to beta blockers
* Severe or uncontrolled asthma or COPD (chronic obstructive pulmonary disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2021-06-17 (Actual)

PRIMARY OUTCOMES:
Identify the correlation between our new RT-qPCR assay for circulating tumor cells and the change in responses in patients on treatment to MRI results. | Baseline, end of cycle 2, end of cycle 4, approximately 6 months depending on treatment plan
  Identify the correlation between our new RT-qPCR assay for circulating tumor cells and the change in responses in patients on treatment to MRI results. We will use 1 to indicate progression of disease seen on brain MRI, 2 to indicate stability or no change in imaging, and 3 to indicate response to treatment. The correlation will be assessed by Spearman's Rank Correlation coefficient. We will have six patients on this study which will give us 12 changed measurements.

SECONDARY OUTCOMES:
Evaluate response with the addition of carvedilol to standard chemotherapy in the second line treatment in glioblastoma multiforme | Baseline, end of cycle 2, end of cycle 4, approximately 6 months depending on treatment plan
  Evaluate response with the addition of carvedilol to standard chemotherapy in the second line treatment in glioblastoma multiforme. Evaluate the correlation between changes in measurements derived from this new assay with changes in a numerical scale based upon brain MRI results. We will use 1 to indicate progression of disease seen on brain MRI, 2 to indicate stability or no change in imaging, and 3 to indicate response to treatment. The correlation will be assessed by Spearman's Rank Correlation coefficient. We will have six patients on this study which will give us 12 changed measurements. We are evaluating the changes of responses in patients on treatment to MRI results and correlate those with our new RT-qPCR assay for circulating tumor cells.
Evaluate incidents of adverse events during the time subjects are taking carvedilol with chemotherapy | From Baseline to 30 days after stopping carvedilol.
  Evaluate adverse events during the time subjects are taking carvedilol with chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Kolodney, MD, Principal Investigator — West Virginia University
Locations (1):
- WVU Cancer Institute - Mary Babb Randolph Cancer Center, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No